CLINICAL TRIAL: NCT05130229
Title: Community Partnership for Healthy Sleep: Sleep Well, Bee Well Part 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000026375; 1R34NR019283-01A1 (NIH)
Record Dates: First submitted 2021-11-16; First posted 2021-11-23 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Pediatric Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Well Bee Well (Experimental): Sleep program to help toddlers sleep better
  Interventions: Behavioral: Sleep Well Bee Well
- Wait-list Control (Placebo Comparator): The wait-listed group will begin the intervention after the intervention group
  Interventions: Behavioral: Sleep Well Bee Well

INTERVENTIONS:
Behavioral: Sleep Well Bee Well — Sleep program to help toddlers sleep better

SUMMARY:
Using a pragmatic cluster randomized trial, this study aims to examine the feasibility, and acceptability of a 3-week behavioral sleep intervention, Sleep Well, Bee Well (SWBW), and to test the preliminary efficacy of SWBW compared to a wait-list control with children ages 1-2.5 years old at two Early Head Start (EHS) centers on toddler sleep characteristics and parent wellbeing.

DETAILED DESCRIPTION:
The first phase of this study is under another study (please see NCT03045874). For this study (Phase II), a pilot pragmatic cluster randomized trial to test the feasibility and preliminary efficacy of SWBW in improving sleep health in children ages 1-2.5 years attending two Early Head Start (EHS) programs will be studied.

A total of 44 families of 1-2.5 year-old healthy children and EHS teachers from both childcare centers will be enrolled. The program teaches early childhood educators about healthy sleep for young children and will train them to be confident facilitators of educational conversations about sleep with parents.

The following specific aims will be addressed with this study: (1) Determine the feasibility of SWBW among 44 families of 1-2.5-year-old healthy children and EHS teachers from both childcare centers; (1a) refine and standardize the SWBW intervention materials (videos, handouts, activities); (1b) determine the feasibility (acceptability, demand, implementation, practicality, adaptation, integration, expansion, and limited-efficacy testing) of the SWBW intervention, study design and recruitment goals; (2) Evaluate the preliminary efficacy of SWBW in 22 intervention and 22 wait-list control parent-child dyads on (2a) toddlers' sleep health (duration, timing, continuity), bedtime routines and parent and EHS teacher sleep knowledge and (2b) toddler's social-emotional health, bedtime routines, parent well-being and parent-teacher engagement. The results from this pilot study will provide support for a future larger-scale cluster-randomized trial that will be fully powered to test the effects of the SWBW program in multiple EHS programs enrolled in the New England Head Start Association.

Parent questionnaires and sleep characteristics of children (actigraphy and parent report) will be collected at three timepoints- Time 1, 2, and 3. Time 1 is the first Baseline Data Collection for the Waitlist Control Group and Intervention Group, and these data will be collected prior to either group starting the 3-week SWBW intervention. Between Time 1 and Time 2, the Intervention Group will receive the 3-week SWBW intervention at the childcare center. Time 2 data collection for both groups will occur during the week following the completion of the intervention received by the Intervention Group. Time 2 data will serve as post-intervention data for the Intervention Group. Time 2 data will also be compared to the first baseline data collected during Time 1 to account for the Waitlist Control Group's waiting time and be used as secondary baseline pre-intervention data for the Waitlist Control Group. Lastly, Time 3 is the Post-Intervention Data Collection for the Waitlist Control Group and will be examined to assess the sustainability of the intervention in the Intervention Group.

ELIGIBILITY:
Inclusion Criteria for parent:

* Primary caregiver of toddler (e.g. mom, dad, aunt, grandparent)
* Fluent in English/Spanish
* Parents of 12-36 month old children

Inclusion Criteria for Toddler:

- Attending either LuLac or West Haven Child Development Center program

Exclusion Criteria for Toddler:

* Diagnosed with sleep apnea
* Travel across 2 or more time zones in the 2 weeks prior to enrollment
* Engaged in concurrent behavioral management for sleep concerns by either primary care providers or sleep specialist.
* Other diagnosed health problem known to be associated with sleep problems (e.g. cerebral palsy, genetic disease, Down's syndrome).

Inclusion / Exclusion Criteria for EHS Teacher:

* Must be over 18 years old
* Speak English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Children's bedtime | 21 days
  The bedtime sleep characteristics will be measured with the Respironics Actiwatch AW2, an accelerometer placed on the toddler's ankle. Reliability for actigraphy in toddlers ranges from .67-.85 when measuring sleep duration. The toddlers will wear the water resistant Actiwatch 2 for seven 24-hour periods at Time 1, 2, and 3. The investigators hypothesize that SWBW will improve toddlers' objectively measured bedtime (goal: bedtime before 9:00PM or at least 45 minutes earlier from baseline). Actigraphs are manually reviewed with sleep diaries for confirmation and scoring of variables is done in Actiware software then processed in R and submitted to statistician for calculation.
Change in Bedtime Variability | 21 days
  Night-to-night variability of bedtime will be calculated using a series of successive differences created by calculating the differences among adjacent observations within the same subject from the Actiwatch 2 data at Time 1, 2, and 3. The mean squared successive differences can be used to compute the MSSD that is considered to be an index of variability/instability. The investigators hypothesize that SWBW will improve toddlers' objectively measured bedtime variability. Actigraphs are manually reviewed with sleep diaries for confirmation and scoring of variables is done in Actiware software then processed in R and submitted to statistician for calculation.
Change in Children's sleep duration | 21 days
  The sleep characteristic of sleep duration will be measured with the Respironics Actiwatch AW2, an accelerometer placed on the ankle of the toddlers. Reliability for actigraphy in toddlers ranges from .67-.85 when measuring sleep duration. The toddler will wear the water resistant Actiwatch 2 for seven 24-hour periods at Time 1, 2, and 3. The investigators hypothesize that toddler's sleep duration will increase by 45 minutes after receiving the SWBW intervention. Actigraphs are manually reviewed with sleep diaries for confirmation and scoring of variables is done in Actiware software then processed in R and submitted to statistician for calculation.
Change in Children's Sleep Duration Variability | 21 days
  Night-to-night variability of sleep duration will be calculated using a series of successive differences created by calculating the differences among adjacent observations within the same subject from the Actiwatch 2 data at Time 1, 2, and 3. The mean squared successive differences can be used to compute the MSSD that is considered to be an index of variability/instability. The investigators hypothesize that SWBW will improve toddlers' objectively measured sleep duration variability. Actigraphs are manually reviewed with sleep diaries for confirmation and scoring of variables is done in Actiware software then processed in R and submitted to statistician for calculation.
Change in Bedtime Routine | 21 days
  Parent reported sleep characteristics will be measured with the Brief Infant Sleep Questionnaire-Revised (BISQ-R) at Time 1, 2, and 3. Each BISQ-R subscale and total score are scaled from 0 to 100. The BISQ-R has been validated against sleep diaries and actigraphy to elicit parent reports of children's sleep patterns (daytime and nocturnal sleep duration, frequency of awakening, sleep latency), sleep habits [sleeping arrangements, parent-child interactions about sleep (e.g., bedtime behaviors, behaviors related to nocturnal awakenings)], sleep difficulty (i.e., bedtime resistance, nocturnal awakenings, and snoring, a risk factor for sleep apnea]. Questions include information about bedtime routine activities and consistency. Approximate time to complete: 10 minutes. The investigators anticipate an improvement in the three subscales and total score of the parent-reported sleep characteristics after receiving the SWBW intervention.
Change in Bedtime Routine | 12 days
  Data on the number of vocalizations and level of noise will be collected using the Language Environment Analysis (LENA) recorder and software that measures frequency of vocalization/verbalizations and conversational turns in children. The LENA device will be worn inside of a vest provided to each child that will be worn on top of the children's clothing. Digital audio recordings will be collected for four days at Time 1, 2, and 3 while the child is wearing the actigraph. Software algorithms parse the continuous audio stream into discrete, variable-length segments that are matched to pre-defined sound models, separating speech-related sounds from environmental and other sounds to compute count estimates of adult words, child vocalizations, conversational turns, and decibel levels.
Change in Children's Bedtime Routine | 21 days
  Parental Interactive Bedtime Behavior Scale (PIBBS) is a 19-item Likert-type parent questionnaire that measures the interactive behaviors caregivers use with their children at bedtime. A total score is calculated as percentage. Approximate time to complete: 5 minutes. The survey will be collected at Time 1, 2, and 3. This survey will be used to generate hypotheses for future clinical trials with a larger sample size. The investigators anticipate that parental interactive bedtime behaviors will improve upon completion of the SWBW intervention.
Change in Parent reported sleep characteristics | 21 days
  Parent reported sleep characteristics will be measured with the Brief Infant Sleep Questionnaire-Revised (BISQ-R) at Time 1, 2, and 3. Each BISQ-R subscale and total score are scaled from 0 to 100. The BISQ-R has been validated against sleep diaries and actigraphy to elicit parent reports of children's sleep patterns (daytime and nocturnal sleep duration, frequency of awakening, sleep latency), sleep habits [sleeping arrangements, parent-child interactions about sleep (e.g., bedtime behaviors, behaviors related to nocturnal awakenings)], sleep difficulty (i.e., bedtime resistance, nocturnal awakenings, and snoring, a risk factor for sleep apnea]. Approximate time to complete: 10 minutes. The investigators anticipate an improvement in the total score of the parent-reported sleep characteristics after receiving the SWBW intervention.

SECONDARY OUTCOMES:
Change in Toddler social-emotional health | 21 days
  SWYC: The Survey of Well-being of Young Children (SWYC)™ is a freely available, simple, comprehensive screening instrument for children under 5 years of age. It requires about 15 minutes to complete. It will be collected at Time 1, 2, and 3. There are 12 aged-based SWYC forms. Every SWYC form includes sections on developmental milestones, behavioral/emotional development, and family risk factors. The investigators anticipate that children will have improved behavioral/emotional development scores after receiving the SWBW intervention.
Change in Parenting stress | 21 days
  The Parenting Stress Index 4-short form (PSI4-SF) is a 36-item parent self-report questionnaire that assesses the level of stress in the parent-child system with a reading level of grade 3.5. It has been well-validated as a measure to predict parenting behavior in the U.S. and more than 20 countries. There are three subscales, parental distress, parent-child dysfunctional interaction, and difficult child, that combine to form a total stress scale Approximate time to complete: 10 minutes. The survey will be collected at Time 1, 2, and 3. The scores range from 36-180. The investigators anticipate that the parenting stress will improve after receiving the SWBW intervention.
Change in Depressive symptoms among parents | 21 days
  The Center for Epidemiological Studies Depression Scale (CES-D) is a brief measure of depressive symptoms that consists of 20 items selected from other depression scales. Each item is rated on a scale from 0-3 in terms of frequency of occurrence during the past week. The total score may range from 0-60, with a score of 16 or more indicating impairment. The reliability of the CES-D has been documented with high internal consistency reliability, acceptable test-retest stability, and construct validity in both clinical and community samples and has been used successfully (alphas = .85-.83) with urban parents. The survey will be collected at Time 1, 2, and 3. The investigators anticipate that the self-report of the parents' depressive symptoms will improve after receiving the SWBW intervention.
Change in Self-report of parental self-efficacy | 21 days
  Self-efficacy for Parenting Tasks Index - Toddler Scale (SEPTI-TS) will be used to measure parental self-efficacy, a key factor in social cognitive theory. The SEPTI-TS is a 51-item questionnaire with seven subscales: emotional competence, sensitive response, protection, discipline/limit setting, play, teaching, and instrumental care/structure/routines. The internal consistency in a study using social cognitive theory to assess parental efficacy in toddlers was good (alpha=0.88). Approximate time to complete: 5 minutes. The survey will be collected at Time 1, 2, and 3. The score ranges from 26-156.The investigators anticipate that parents will report increased parental self-efficacy upon completion of SWBW.
Change in Parental knowledge and beliefs about children's sleep | 21 days
  Knowledge, attitudes, self-efficacy, and beliefs about sleep in children (KASB) will be administered. There are seven self-efficacy items. The survey will be collected at Time 1, 2, and 3. The score ranges from 0-76. The investigators anticipate that parental knowledge, attitudes, self-efficacy, and beliefs about their children's sleep will improve upon completion of the SWBW intervention.

OTHER OUTCOMES:
Intervention feasibility and acceptability | 21 days
  To determine the feasibility and acceptability of SWBW among families of 12-30-month-old healthy toddlers and EHS teachers, data will be collected using study-specific Likert-scale surveys. Biweekly site visits and recorded field notes on fidelity will be collected. Together, these field notes will assist in determining the need for intervention refinement and standardization of the intervention manual in preparation for a larger, full-scale future trial.
  The feasibility goals include >50% enrollment and >80% retention rates based on published physical activity and obesity intervention research in Head Start preschool programs. Approximate time to complete: 10 minutes. This will be collected at the end of the intervention. The investigators anticipate that the program will be acceptable and feasible to the EHS centers, teachers, and parents.
Children's nap timing | 21 days
  The sleep characteristic of nap timing will be measured with the Respironics Actiwatch AW2, an accelerometer placed on the toddler's ankle. Reliability for actigraphy in toddlers ranges from .67-.85 when measuring sleep duration. The toddler will wear the water resistant Actiwatch 2 for seven 24-hour periods at Time 1, 2, and 3. The investigators hypothesize that toddlers' day-to-day nap variability will be reduced after receiving the SWBW intervention.
Change in Self-report of parents' sleep disturbance | 21 days
  PROMIS- Parent Sleep short form is a 7-item survey developed from the item bank of the Patient-Reported Outcomes Measurement Information System (PROMIS™) Sleep Disturbance (SD) to identify sleep disturbance in adults. The survey will be completed at Time 1, 2, and 3. The score ranges from 8-40. The investigators anticipate that parents' self-report of sleep disturbances will improve upon completion of the SWBW intervention.
Change in Self-report of parents' hopefulness | 21 days
  Future/Hope Scale: The 12-item Trait Hope Scale (also referred to as The Future Scale) assesses hopefulness. It has two subscales: Pathways and Agency. It has a Cronbach's alpha of between .74 to .84, depending on the population. The Cronbach's alpha for the Agency subscale is between .71 to .76, and between .63 to .80 for the Pathways subscale. The survey will be collected at Time 1, 2, and 3. The score ranges from 8-64. The investigators anticipate that parents will report increased hopefulness upon completion of SWBW.
Sleep Diary | 21 days
  Parents will complete a sleep diary to record their toddler's naptime, bedtime, duration of sleep, sleep location, and bedsharing for the 7-day period when the toddlers wear the Actiwatch 2 (see below). These data will assist with the actigraphy scoring. The sleep diary will be collected at Time 1, 2, and 3.
Change in Parental Physical and Mental Health | 21 days
  SF-36 (general physical and mental health): The SF-36 is a multi-purpose survey designed to capture adult patients' perceptions of their own health and well-being. Based on a much longer survey developed in the 1980's by Ware, J.E., the SF-36 has 36 items grouped in 8 dimensions: physical functioning, physical and emotional limitations, social functioning, bodily pain, general and mental health. It is a generic measure, as opposed to one that targets a specific age, disease, or treatment group. In one of the first validity studies, the instrument was acceptable to good estimates of reliability, support for construct validity, and support for convergent and divergent validity for 4 of the 8 dimensions. The survey will be collected at Time 1, 2, and 3. The score ranges from 0-100. The investigators anticipate that the parents' self-report of their well-being will improve upon completion of the SWBW intervention.
Change in Parent-Teacher Involvement | 21 days
  We will measure the quality of parent-teacher interaction using the INVOLVE questionnaires with both the EHS teachers and parents. The 11-item parent-reported Parent-Teacher Involvement Questionnaire (INVOLVE-P) was adapted for use with parents of children in Head Start programs to evaluate parents' involvement with their children's education and activities at home and at childcare. As a companion measure, the 20-item teacher-reported Parent-Teacher Involvement Questionnaire (INVOLVE-T) requires teachers to rate parents' involvement in their child's education, and their frequency of contact with teachers and school personnel. There are three subscales were created: Teacher Bonding with Parent, Parent Involvement in Education, and Parent Involvement with Teacher. These surveys will be collected at Time 1, 2, and 3. The range of scores for the INVOLVE-P is 0-104; the range of scores for the INVOLVE-T is 0-80.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Ordway, PhD, Principal Investigator — Associate Professor of Nursing
Locations (2):
- United States (2):
  - Lulac Head Start, Inc., New Haven, Connecticut
  - West Haven Child Development Center, West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No